CLINICAL TRIAL: NCT01342822
Title: A Prospective, Randomized, Multi-center Trial to Assess the Everolimus-Eluting Coronary Stent System (PROMUS Element) for Coronary Revascularization in a Population of Unrestricted Patients
Brief Title: Trial to Assess the Everolimus-Eluting Coronary Stent System (PROMUS Element) for Coronary Revascularization
Acronym: PLATINUM+
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: BSI-01
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Ischemic Heart Disease; Coronary Artery Stenosis
Keywords: Heart disease; Coronary Revascularization
MeSH Terms: conditions — Myocardial Ischemia; Coronary Stenosis; Heart Diseases | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PROMUS Element™: All patients enrolled will be randomized 2:1 to receive the PROMUS Element™ stent (N=1987)
  Interventions: Device: Angioplasty (PROMUS Element™, and Xience™ Prime stent)
- Xience™ Prime stent: All patients enrolled will be randomized 2:1 to receive the PROMUS Element™ stent (N=1987) versus the Xience™ Prime Stent (N=993).
  Interventions: Device: Angioplasty (PROMUS Element™, and Xience™ Prime stent)

INTERVENTIONS:
Device: Angioplasty (PROMUS Element™, and Xience™ Prime stent) — Patients with symptomatic ischemic heart disease due to stenotic lesions amenable to percutaneous treatment with a drug eluting stent in a consecutive unselected patient population, provided that the proposed research use of the product is consistent with the approved (labeled) uses of such product and with the reimbursed indications (in countries where reimbursement procedure applies, eg France) and does not violate any other applicable law, regulation or ethical directive/code.

SUMMARY:
The PROMUS Element™ clinical trial (PLATINUM-PLUS) consists of a randomized controlled trial (RCT) in the European Union (EU) which will enroll approximately 2980 subjects (2:1 randomization PROMUS Element™: Xience™ Prime) in a Population of consecutive, all comers in the reimbursed indications per-country

All subjects will be screened per the protocol required inclusion/exclusion criteria.

DETAILED DESCRIPTION:
The PLATINUM-PLUS trial will investigate in a broad patient and lesion population, the CE Mark approved PROMUS Element™ Everolimus-Eluting Coronary Stent System (PROMUS Element), which combines the Element™ stent (the latest generation stent from Boston Scientific Corporation [BSC, Natick, Massachusetts, United States]), everolimus, and the poly (n butyl methacrylate) (PBMA) and poly (vinylidene fluoride co hexafluoropropylene) (PVDF-HFP) polymers. The PROMUS Element, received CE Mark on November 3rd 2009; it is currently under investigation in the PLATINUM clinical trial, and has great promise as it combines BSC's novel stent technology with the everolimus drug and polymers that have demonstrated excellent performance in the SPIRIT clinical program.

PROMUS Element comprises the following key components: everolimus, 2 polymers, and the Element stent component. The same everolimus and polymer combination is commercially available in many countries on the MULTI-LINK VISION™ stent. It is manufactured and distributed by Abbott as the XIENCE™ V Everolimus Eluting Coronary Stent System (XIENCE V), and also distributed by BSC as the identical stent system, also manufactured by Abbott, as the PROMUS™ Everolimus-Eluting Coronary Stent System (PROMUS). The names XIENCE V and PROMUS are used synonymously within this protocol.

While PROMUS Element is a new DES system, its constituent parts are either approved by the Food and Drug Administration (FDA, i.e., drug and polymers from PROMUS, P070015), are under investigation in an FDA-approved trial (i.e., Element stent component in the PERSEUS trial, G060237), or have received an approvable letter from the FDA. The balloon component material of the PROMUS Element delivery system is the same as that used in TAXUS Liberté (P060008), which received an approvable letter on February 11, 2008. The PROMUS Element stent delivery system is from the Apex™ Monorail™ PTCA Dilatation Catheter (P860019/S208), which received an approvable letter on October 24, 2006. Table 1 compares the TAXUS Express2, TAXUS Liberté, and PROMUS Element stent systems.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. The patient must be ≥18 of age
2. Symptomatic ischemic heart disease (CCS class 1-4, Braunwald Class IB, IC, and/or objective evidence of myocardial ischemia);
3. Acceptable candidate for CABG;
4. The patient is willing to comply with specified follow-up evaluations;
5. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics Committee (MEC).

   Angiographic Inclusion criteria:
6. Single or multiple native coronary artery or saphenous vein graft lesions in single or multiple vessels;
7. Patients with multi-lesion or multi-vessel coronary disease may undergo staged (planned) procedures within 30-days of the index procedure.
8. Reference vessel diameter must be ≥2.25 to ≤ 4.25 mm by visual estimate.

Exclusion Criteria:

1. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test;
2. Patients in whom anti-platelet and/or anticoagulant therapy is contraindicated;
3. Patient has other medical illness (e.g., cancer, known malignancy , congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year);
4. Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, prasugrel, platinum chromium alloy, everolimus, and/or contrast sensitivity that cannot be adequately pre-medicated;
5. Patient with LVEF <20%, cardiogenic shock, or hemodynamic compromise requiring pressors or inotropes or mechanical support devices
6. Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
7. Currently participating in another investigational drug or device study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comers, in the indications reimbursed in the participating countries
Sampling Method: Non-Probability Sample
Enrollment: 2980 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Target Vessel failure (TVF) | 12 months
  Target Vessel failure (TVF) of the PROMUS Element™ Everolimus-Eluting Coronary Stent at 12 months post-procedure. TVF is defined as any ischemia-driven revascularization of the target Vessel (TVR), MI (Q-wave and non-Q-wave) related to the target vessel, or cardiac death related to the target vessel.

SECONDARY OUTCOMES:
Clinical endpoints | 30 days, 12 months and 24 months
  Ischemia Driven TLR and TVR rate, TLF rate: defined as any ischemia-driven TLR, MI (Q-wave and non-Q-wave)related to the target vessel, or cardiac death related to the target vessel MI rate: Q-wave and non-Q-wave, cumulative and individual, Cardiac death rate, Non-cardiac death rate, All death or MI rate All Death/MI/TVR rate, MACE rate defined as a composite of death, MI (Q wave or non-Q wave), emergent CABG, or TLR by repeat PTCA or CABG. Stent Thrombosis (ST)rate.

CONTACTS AND LOCATIONS:
Locations (50):
- France (19):
  - Clinique de l'Europe, Amiens
  - Polyclinique de Bois Bernard, Bois-Bernard
  - Clinique Saint Augustin, Bordeaux
  - CHU Brest, Brest
  - Clinique Saint-Martin, Caen
  - CHG Chartres, Chartres
  - CHU Grenoble, Grenoble
  - CH Lagny, Lagny
  - Hôpital privé Beauregard, Marseille
  - Institut Hospitalier Jacques Cartier - ICPS, Massy
  - Clinique les Fontaines, Melun
  - Clinique du Millénaire, Montpellier
  - Nouvelles Cliniques Nantaises NCN, Nantes
  - Hôpital Privé Les Franciscaines, Nîmes
  - Clinique Saint-Pierre, Perpignan
  - Centre Privé Claude Galien, Quincy-sous-Sénart
  - Groupement de Coopération Sanitaire, Saint-Nazaire
  - Clinique Pasteur, Toulouse
  - CHU Rangueil, Toulouse
- Germany (4):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Klinikum Leverkusen, Leverkusen
  - Kardiologische Praxis und Praxisklinik, München
  - Universitätsklinikum Ulm, Ulm
- Italy (7):
  - Azienda Ospedale "S.G. Moscati", Avellino
  - Ospedale Civile di Legnano, Legnano
  - Ospedale Carlo Poma, Mantova
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero-Universitaria Pisana - MCV I°, Pisa
  - Azienda Ospedaliera "Ordine Mauriziano di Torino", Torino
  - Azienda ULSS 9 Treviso; Ospedale "S. Maria di Ca' Foncello", Treviso
- Albert Schweitzer Ziekenhuis, Dordrecht, Netherlands
- University Clinic of Cardiology, Skopje, North Macedonia
- Spain (10):
  - Hospital General Yague, Burgos, Spain
  - Hospital Infanta Cristina, Badajoz
  - Hospital German Trias i Pujol, Badalona
  - Hospital Sant Pau i Sant Creu, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Valdecilla, Santander
  - Hospital del Mexoeiro, Vigo
- University Hospital Fribourg, Fribourg, Switzerland
- United Kingdom (7):
  - Royal Victoria Hospital, Belfast
  - Lancashire Cardiac Centre, Blackpool
  - Royal Sussex County Hospital, Brighton
  - St Thomas Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Craigavon Cardiac Centre, Portadown
  - Royal Victoria Hospital, Wolverhampton